CLINICAL TRIAL: NCT07310407
Title: Evaluation of the Effect of Rutin and Vitamin C in Patients With Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD)
Brief Title: Rutin and Vitamin C in Patients With Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaimaa salem, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC Approval Number: REC # 414
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Rutin; Ascorbic Acid; Diet; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ruta C group (Experimental): Drug: Rutin + Vitamin C - Oral, two tablets containing 60 mg Rutin + 160 mg Vitamin C, three times daily for 12 weeks, plus lifestyle intervention (Mediterranean diet and structured exercise).
  Interventions: Drug: Rutin + Vitamin C
- Vitamin C group (Experimental): Drug: Vitamin C - Oral capsules, 500 mg, twice daily for 12 weeks, plus lifestyle intervention (Mediterranean diet and structured exercise).
  Interventions: Drug: Vitamin C 500mg
- Control group (Experimental): Behavioral: Lifestyle Intervention - Mediterranean diet focusing on fruits, vegetables, whole grains, healthy fats, and structured exercise program for 12 weeks
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Drug: Rutin + Vitamin C — Type: Drug (Combination therapy) Details: Oral administration of two tablets containing 60 mg Rutin + 160 mg Vitamin C, taken three times daily for 12 weeks.
  Other Names: Ruta C
  Arms: Ruta C group
Drug: Vitamin C 500mg — Type: Drug (Single agent) Oral administration of Vitamin C 500 mg, taken twice daily for 12 weeks
  Other Names: C-Retard
  Arms: Vitamin C group
Behavioral: Lifestyle Intervention — Mediterranean diet focusing on fruits, vegetables, whole grains, healthy fats, plus structured exercise program for 12 weeks.
  Other Names: diet and exercise
  Arms: Control group

SUMMARY:
evaluate the combined effects of Rutin and Vitamin C versus Vitamin C alone on selected oxidative stress markers, inflammation, hepatic steatosis regression, and associated metabolic parameters in patients with MASLD

DETAILED DESCRIPTION:
Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) is a common liver disorder with risks of progression to fibrosis, cirrhosis, and hepatocellular carcinoma.

Its global prevalence is high, driven by oxidative stress and impaired antioxidant defenses, while no approved pharmacological treatments currently exist. Nutritional agents such as vitamin C and rutin show promise in improving liver function and reducing oxidative damage.

This study will evaluate their combined effects in addressing MASLD's multifactorial pathology.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Metabolic-Associated Steatotic Liver Disease (MASLD).

Exclusion Criteria:

* HCV infection.
* HBV infection.
* Patients with a history of significant alcohol consumption.
* Autoimmune hepatitis.
* Celiac disease (CD).
* Wilson's disease (WD).
* Haemochromatosis.
* Drugs: Tamoxifen, Valproic acid, Amiodarone, Methotrexate, steroids and immunosuppressive agents, oral contraceptive pills, or drugs that can affect liver profile.
* Hypo or hyper thyroidism.
* Bypass surgeries.
* TPN (Total Parenteral Nutrition).
* Pregnant individuals or patients planning to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
• Change in tumor necrosis factor-alpha (TNF-α) levels from baseline to week 12. | 12 weeks
  Serum TNF-α, a key biomarker of inflammation in MASLD

SECONDARY OUTCOMES:
• Change in serum malondialdehyde (MDA) levels from baseline to week 12. | 12 weeks
  Malondialdehyde (MDA) is a well-established biomarker of oxidative stress in MASLD, reflecting lipid peroxidation and liver injury.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Zaki, Professor, Study Director — Ain Shams University
Locations (1):
- National Hepatology and Tropical Medicine Research Institute (NHTMRI), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No